CLINICAL TRIAL: NCT06389396
Title: Investigation of a New Rectal Catheter for Users of Transanal Irrigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP362
Record Dates: First submitted 2024-04-11; First posted 2024-04-29 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Bowel Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device - newly developed TAI catheter. (Experimental): CP362 Test Catheter: The investigational device is intended to perform TAI procedures together with the CE-marked Peristeen® Plus TAI system.
  Interventions: Device: CP362 Test Catheter
- Peristeen Plus (No Intervention): Comparator catheter: The Peristeen® Plus rectal balloon catheter is used together with the CE-marked Peristeen® Plus TAI system.

INTERVENTIONS:
Device: CP362 Test Catheter — The investigational device is intended to perform TAI procedures together with the CE-marked Peristeen Plus TAI system.
  Arms: Investigational device - newly developed TAI catheter.

SUMMARY:
The clinical investigation is an exploratory, randomised controlled, open-labelled, crossover investigation.

The clinical investigation will be conducted as a multi-centre clinical investigation in two different clinical investigation sites in Denmark.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written Informed Consent
2. Is at least 18 years old
3. Has full legal capacity
4. Has used Trans Anal Irrigation (TAI) with balloon catheter for at least 4 weeks prior to inclusion
5. Performs TAI minimum 3 times/week
6. Is able to follow study procedures assessed by investigator

Exclusion Criteria:

1. Has known anal or colorectal stenosis
2. Has active/recurrent colorectal cancer
3. Is within 3 months of anal or colorectal surgery
4. Is within 4 weeks of endoscopic polypectomy
5. Has ischaemic colitis
6. Has acute inflammatory bowel disease
7. Has acute diverticulitis
8. Is participating in any other clinical study that may interfere with this study (assessed by investigator).
9. Is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Århus Universitetshospital, Aarhus, Jutland
  - Amager Hvidovre Hospital, Hvidovre, Region Sjælland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2024 and July 2024, 20 users were recruited for the study from two sites and encompassed the Intention to treat (ITT) population.
Pre-assignment Details: The 20 recruited participants were randomized into the two intervention arms. No participants were excluded or discontinued. No adverse events were reported.
Groups:
- Investigational Device Then Comparator Device: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 4.
  At the first intervention the transanal irrigation (TAI) procedure was performed with the CP362 Test Catheter together with the CE-marked Peristeen® Plus TAI system, then, at the second intervention the TAI procedure was performed with the Comparator catheter, the Peristeen® Plus rectal balloon catheter, together with the CE-marked Peristeen® Plus TAI system.
- Comparator Device Then Investigational Device: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 4.
  At the first intervention the transanal irrigation (TAI) procedure was performed with the Comparator catheter, the Peristeen® Plus rectal balloon catheter, together with the CE-marked Peristeen® Plus TAI system, then, at the second intervention the TAI procedure was performed with CP362 Test Catheter together with the CE-marked Peristeen® Plus TAI system
Period: Visit 1
Arm/Group | Investigational Device Then Comparator Device | Comparator Device Then Investigational Device
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | Investigational Device Then Comparator Device | Comparator Device Then Investigational Device
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- Total ITT Population: Each investigation arm consisted of two test visits. On each visit, the participants underwent one TAI procedure with either the CP362 test catheter or the Comparator catheter, according to the randomization scheme.
Arm/Group | Total ITT Population
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 20

OUTCOME MEASURES:

1. Primary Outcome: Was it Possible to Perform Transanal Irrigation?
Description: After visit 1 and visit 2, the primary endpoint, defined as if it was possible to perform transanal irrigation, was answered by a yes/no answer.
Time Frame: Evaluated at Visit 1 and Visit 2 (within a time duration of up to 17 days)
Population: The full analysis set
Measure: Number; unit: Number of participants who replied YES
Groups:
- Investigational Device - Newly Developed TAI Catheter.: The CP362 Test Catheter, the investigational device, was used to perform TAI procedures together with the CE-marked Peristeen® Plus TAI system.
- Comparator Device - Peristeen Plus: Comparator catheter. The Peristeen® Plus rectal balloon catheter, was used together with the CE-marked Peristeen® Plus TAI system.
Arm/Group | Investigational Device - Newly Developed TAI Catheter. | Comparator Device - Peristeen Plus
Number analyzed (Participants) | 20 | 20
Number of participants who replied YES | 20 | 20

ADVERSE EVENTS:
Time Frame: Adverse events were registered from the individual's enrolment until termination in the study. The total study duration for the individual subject was between two to 17 days, consisting of three site visits (V0-V2), where V0 and V1 could be performed the same day.
Description: [Not specified]
Groups:
- Comparator Catheter - Peristeen Plus: Comparator catheter: The Peristeen® Plus rectal balloon catheter is used together with the CE-marked Peristeen® Plus TAI system.
Arm/Group | Investigational Device - Newly Developed TAI Catheter. | Comparator Catheter - Peristeen Plus
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT06389396/Prot_SAP_000.pdf